CLINICAL TRIAL: NCT00631735
Title: Perceptions of Touch in People With Cancer
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Kalman, RN, PhD, SUNY UMU
Other Study IDs: 5452
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Cancer
Keywords: cancer; qualitative
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is a qualitative, phenomenological research design. The research question is the lived experience of adult oncology patients undergoing chemotherapy being touched and touching. The researcher will conduct minimally-structured interviews with a set of follow-up interviews to verify interpretations and ascertain additional participant reflections on the phenomenon of touch. The purpose of this study is to describe the sensation of touch in adult oncology patients who are actively undergoing chemotherapy treatment. The primary objective is to identify the essences of multiple meanings of touch to these patients. The importance of touch in physiological development, learning patterns, and stress reduction has been demonstrated in humans and animals through years of research (Field, 2000). Based on research which indicates touch therapies provide a significant amount of symptom relief and reduction in anxiety, a growing number of hospitals and clinics are integrating massage therapy into services provided to patients in order to ameliorate many symptoms of diagnosis and/or treatment-related discomfort. Examples are the integrative medicine programs at Memorial Sloan-Kettering Cancer Center and George Washington University Medical Center which include touch therapy modalities. Research focusing on the embodied experience of sensory phenomena such as touch is important to provide the basis for more effective care. No studies to date have focused on the self-reported experience of the cancer patient with regard to what touch means to these individuals, particularly those actively in treatment with intravenous chemotherapy. The embodied sensation of touch in these people is important to understand in order to provide more effective touch-based interventions and also to increase awareness of direct care staff, including nurses, of the profound and complex effect that all forms of touch have on those who are physically and psychically vulnerable.

DETAILED DESCRIPTION:
The importance of touch in physiological development, learning patterns, and stress reduction has been demonstrated in humans and animals through years of research. Based on research which indicates touch therapies provide a significant amount of symptom relief and reduction in anxiety, a growing number of hospitals and clinics are integrating massage therapy into services provided to patients in order to ameliorate many symptoms of diagnosis and/or treatment-related discomfort. Examples are the integrative medicine programs at Memorial Sloan-Kettering Cancer Center and George Washington University Medical Center which include touch therapy modalities. Research focusing on the embodied experience of sensory phenomena such as touch is important to provide the basis for more effective care. No studies to date have focused on the self-reported experience of the cancer patient with regard to what touch means to these individuals, particularly those actively in treatment with intravenous chemotherapy. The embodied sensation of touch in these people is important to understand in order to provide more effective touch-based interventions and also to increase awareness of direct care staff, including nurses, of the profound and complex effect that all forms of touch have on those who are physically and psychically vulnerable. The stress of the diagnosis and treatment heightens patients' awareness of many taken-for-granted aspects of daily interaction, including touching and being touched. The side effects of certain chemotherapy treatments can create neuropathies that make the sense of touch diminished or painful, even to the extent that putting on socks and shoes or taking a pulse or blood pressure can become excruciatingly painful experiences. By allowing people who are actively undergoing treatment for cancer to express the meaning of touch in their lives, a fuller understanding of the multiple dimensions of the experience can be achieved. Using this understanding, more effective nursing and touch interventions can be designed to enhance patient comfort. One author notes a multitude of terminologies to distinguish types of nursing touch in her literature review. She observes that, "it is possible that touch is so integral … that the need for serious research is not recognized … it is clear that more research, and qualitative research in particular, is needed to better understand the effects and meaning of touch…" (p. 849). Chang (2001) stresses the need to treat physical touch in a "holistic way" (p. 821) to positively impact the patient. She also stresses the meaning of physical touch is "dependent on reciprocal expectations about touch," (p.826). Based on the importance of Chang's delineation of multidimensional aspects of perceptions of touch and the mutual nature of the expectations, additional study is warranted to elucidate the perceptions of touch in patients. This understanding can be used to facilitate increased quality of life in patients with cancer through better education of health care providers and integration of complementary modalities in a safe, effective plan of comprehensive care.

The research design will be a phenomenological qualitative design. The purpose of phenomenological research is the description of the experiential meanings we live as we live them. The research question is the lived experience of adult oncology patients undergoing chemotherapy being touched and touching. The researcher will conduct minimally-structured interviews with a set of follow-up interviews to verify interpretations and ascertain additional participant reflections on the phenomenon of touch.

Data will consist of participant interviews recorded and transcribed by the researcher. Following the methodology of Colaizzi (1978), the interviews are read multiple times to immerse the researcher in each participant's text and achieve a collective impression or feeling for the whole. Following this, significant statements are selected from each interview which pertain to the phenomenon under investigation. Meanings of these statements are formulated hermeneutically (i.e., interpreted) by the researcher. These meanings are then grouped according to themes identified by the researcher. All meanings must be considered. An exhaustive description of the phenomenon under investigation is then written which focuses on the universal, essence that lies on the other side of the concreteness of lived meaning. The researcher then returns to the participants for validation of the meanings, clusters, and descriptions. Finally, new data obtained from participants are incorporated into the structure of the research. Prior to conducting interviews and throughout the entire research process, a log is kept of the researcher's presuppositions about the investigated topic. This acknowledgement of the researcher's viewpoint assists in setting these pre-conceived ideas aside in order to come to direct terms and meanings as lived by the participants. One author's contribution to the methodology comes in his approach to the interpretations of the text. He describes the following components of phenomenological interpretation: 1. turning to the nature of lived experience, 2. investigating the lived experience, 3. hermeneutical phenomenological reflection, 4. hermeneutical phenomenological writing, 5. maintaining a strong and oriented relation, and 6. balancing the research context by considering parts and whole. These interpretive relationships are not linear steps; they form a guideline for all phenomenological reflection and writing.

While the concepts of reliability and validity can not be applied to phenomenological research as they are for quantitative studies, the data trail and decisions regarding interpretation are to be documented fully so that thought processes in the identification of essential themes and meanings can be audited by outside reviewers. Trustworthiness of the data and interpretations is paramount in qualitative inquiry. Lincoln and Guba (1985) set forth four basic concepts to establish trustworthiness: truth value, applicability, consistency, and neutrality. They discuss the divergence of the naturalistic paradigm of qualitative research methods from the traditional or positivist paradigm of cause and effect. The four concepts take on the following respective characteristics: credibility, transferability (which requires contextual similarity), dependability, and confirmability.

The first step of the study is the researcher's articulation of presuppositions regarding the phenomenon of touch. This is carried out throughout the process of the study to ensure the process of interpreting and defining essences of participants' experiences are not unduly influenced by the experience of the researcher. Following approval from the Institutional Review Board, participants will be recruited from physician, nurse practitioner, and physician assistant recommendations at the Regional Oncology Center and other central New York oncology clinics. Each patient will be asked by his or her practitioner if he or she wishes to take part in the study. If the person is interested, his or her phone number will be forwarded to the researcher by the practitioner. The researcher will then contact the patient to confirm his or her willingness to participate and understanding of the aims and procedures of the study. For each patient who is confirmed as desiring participation, the researcher will obtain informed written consent. Participants may withdraw at any time during this study until the interview is transcribed, in order to maintain the integrity of the study. All potential physical, social, legal, and other risks will be described and a phone number given to the participants to contact the researchers in case of questions. Each participant will be interviewed for approximately one hour in a private place and at a time which is convenient to the participant and researcher. Before beginning the interview, the participant will be asked to choose a pseudonym. A second interview will take place several months later (after the researcher has had sufficient time to fully immerse herself in the data). This will give the participants a chance to reflect on their interview and review interpretations of their information made by the researcher. Each interview will be taped and field notes taken by the researcher. These will be transcribed soon after the interview to allow initial impressions to be noted along with interview text. Subjects will be enrolled until saturation is reached (no new data obtained from initial interviews). Due to the need for saturation, the number of interviews can not be planned beforehand; however, the number is estimated to be between 8 and 12 participants. The interviews will be transcribed by the researcher or other transcriptionist. To protect confidentiality, the participants' names will not be attached to electronic or paper data; only pseudonyms will be used as interview and data identifiers. All data will be stored in a locked file container accessible only to the researchers. All audiotapes will be destroyed after completion of the research study. The confidentiality agreements will be kept securely in a separate, locked file cabinet also accessible only to the researchers. Participants' demographic information, including age, gender, ethnicity, educational level, and employment (current or before illness) will be collected and stored with the pseudonym.

Interviews will consist of broad open-ended questions. In order to establish rapport and provide a foundation for more detailed questions, the initial questions will begin with the experience of discovering the cancer, diagnosis, the experiences of treatment, and social and personal consequences of the lived experience. Exploration of the initial diagnosis is important because of the life-changing nature of the diagnosis and the accompanying feeling of shock that many people experience at the moment of receiving the diagnosis (American Cancer Society, 2006). The questioning will then focus on the experience of being touched by others, first during the process of the diagnosis and treatment, then prior to this experience. Questions will also be formulated during the interview on the sensation of touch now and prior to treatment, including touching others. All questions will be broad to allow the greatest possible latitude of participant interpretation; however, a general list of questions will be formulated to ensure consistency and completeness of data collection across participants. In general, the interview is paramount in data collection because it is the intention of the researcher to be "minimally intrusive" while eliciting descriptions that are robust and complete in describing each person's perspective of the phenomenon. In this study, several broad questions will be asked at some point during each interview to ensure that similar baseline data are collected for each participant. Questions to be asked will be:

* Please tell me about some of the changes you have experienced since being diagnosed with cancer.
* Please tell me about how you have coped with the diagnosis and treatments.
* How have people around you reacted to your diagnosis?
* How important to you is being touched?
* Has your sense of touch changed in any way since you started chemotherapy?
* Has the amount of physical contact you have with others changed?
* Have you ever had any massage or other form of touch therapy?
* Please describe how it feels to be touched when you are going to the medical clinic or having procedures such as CT scans done.

ELIGIBILITY:
Inclusion Criteria:

* Adults, at least 18 years old, who have been diagnosed with cancer (any form) and are in active treatment.
* Treatment must include intravenous chemotherapy (either as an outpatient or an inpatient) with or without surgery and/or radiation.
* Each participant will be fluent in English, able to hear and speak, fully alert and oriented, able to verbalize both concrete and abstract ideas, and able to comprehend and sign consent for participation.

Exclusion Criteria:

* Anyone else

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults, at least 18 years old, who have been diagnosed with cancer (any form) and are in active treatment. Treatment must include intravenous chemotherapy (either as an outpatient or an inpatient) with or without surgery and/or radiation. Each participant will be fluent in English, able to hear and speak, fully alert and oriented, able to verbalize both concrete and abstract ideas, and able to comprehend and sign consent for participation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The primary objective is to identify the essences of multiple meanings of touch to these patients. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Kalman, RN PhD, Principal Investigator — SUNY UMU
Locations (1):
- SUNY UMU, Syracuse, New York, United States